CLINICAL TRIAL: NCT04407351
Title: Develop Phototherapy of Improving the Quality of Sleep and Healthcare for Patients With Sleep Disorder, Mild Cognitive Impairment, or Dementia: a Novel Light Emitting Diode (LED) Application on Health Promotion
Brief Title: Develop Novel Phototherapy for Health Care of Patients With Sleep Disorder, Mild Cognitive Impairment, or Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Hsin-Su Yu, Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MOST106-3111-Y-043001
Record Dates: First submitted 2020-05-10; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Dementia; Sleep Disorder; Mild Cognitive Impairment; Phototherapy
Keywords: Dementia; Sleep Disorder; Phototherapy; Light Emitting Diode (LED); Mild Cognitive Impairment
MeSH Terms: conditions — Dementia; Sleep Wake Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Green LED light - Red LED light (Other): Every morning between 7-8 o'clock, participants will receive 7,500 Lux at home at 470 nm as a full-band (bright light) light-emitting diode (Green LED light) luminaire with a distance of 80-100 cm at a 45-degree angle Light exposure for 30-60 minutes for 12 weeks, the rest of the time indoors is not limited by light. Then crossover to red light after 2 weeks for wash out. Every morning between 7-8 o'clock, participants receive 50 Lux of Red LED light (dim light) at their own homes and illuminate at a distance of 80-100 cm at a 45-degree angle for 30-60 minutes for 12 weeks.
  Interventions: Device: Green LED light; Device: Red LED light (placebo)
- Arm Red LED light - Green LED light (Other): Every morning between 7-8 o'clock, participants receive 50 Lux of Red LED light (dim light) at their own homes and illuminate at a distance of 80-100 cm at a 45-degree angle for 30-60 minutes for 12 weeks, and the rest of the time indoors is not restricted by light. Then crossover to green light after 2 weeks for wash out. Every morning between 7-8 o'clock, participants will receive 7,500 Lux at home at 470 nm as a full-band (bright light) light-emitting diode (Green LED light) luminaire with a distance of 80-100 cm at a 45-degree angle Light exposure for 30-60 minutes for 12 weeks.
  Interventions: Device: Green LED light; Device: Red LED light (placebo)

INTERVENTIONS:
Device: Green LED light — Investigators arrange 12 weeks green LED light phototherapy.
Device: Red LED light (placebo) — Investigators arrange 12 weeks red LED light phototherapy (placebo).

SUMMARY:
Investigators aim to collaborate with the division of neurology, ophthalmology and dermatology at the Kaohsiung Medical University, and make a new phototherapy for participants suffering from dementia, sleep disorder, mild cognitive dysfunction by using IoT and data science on big health and environmental data.

DETAILED DESCRIPTION:
Solar light is an important environmental factor for all living organisms. With the advancement of the lighting technology, artificial light, such as light emitting diode (LED), has become another major lighting source. The influence of blue light and color temperature emitted from LED light source in most of the commercial 3C electronics on human health has been increasingly paid attention. Light exposure has been reported to be associated with different physiological mechanisms and pathologic events, including sleeping, metabolism and brain dysfunctions. However, lights are also applied in many therapeutic processes. Hence, it is a critical issue to develop a next-generation lighting environment for health promotion and improve the competitiveness of green-technology industries in Taiwan by integrating biomedical researches and cutting-edge lighting technology. For developing next-generation LED industry, the inspection technology and product standard on photobiology safety has been established in Taiwan. Inspiringly, Researchers in Taiwan have made a LED structure that can emit all the hues of sunlight by changing its terminal voltage, which may further facilitate the use of future lighting device on health promotion. Based on these technical advancement, in this project, investigators aim to integrate multidisciplinary investigations on animal experiments, translational applications, and clinical trials to establish an good lighting environment for participants with dementia and mild cognitive dysfunction, and bring benefits to Taiwan's green technologies. To meet this goal, this project aims to integrate lighting and information technologies, including Internet of Things (IoT) and data science analytics, to investigate the lighting effects on human health by conducting animal and translational experiments, and further promote the health in multiple testing groups across different patients. In this project, investigators incorporate the research strengths in light bioscience, environmental bioscience and medical engineering developed at National Health Research Institutes (NHRI) and the lighting, IoT and data science technologies developed at National Applied Research Laboratories (NARL). Additionally, investigators aim to collaborate with the division of neurology, ophthalmology and dermatology at the Kaohsiung Medical University, and make a new phototherapy for participants suffering from dementia, sleep disorder, cognitive dysfunction by using IoT and data science on big health and environmental data. By integrating multi-disciplinary technologies, investigators aim to promote health on brain, mind and body for elderly people and susceptible population by providing a health home lighting environment, which would be potentially beneficial to resolve the emerging issues of aging, sub-health population, psychiatric and neurodegenerative diseases. Moreover, the safety and molecular mechanism of phototherapy will be validated using animal models. Industrially, this project will build a strong linkage between LED, information and health promotion industries and upgrade the traditional LED industry by adding the novel application on health promotion.

ELIGIBILITY:
Inclusion Criteria:

* (1) The age is between 55 and 80 years old
* (2) Education level is above elementary school graduation
* (3) Use Edinburgh Inventory as the right hand

Exclusion Criteria:

* (1) Neurological diseases, including cerebral stroke, epilepsy, Parkinson's disease and head trauma that cause local nerve signs
* (2) Mental illnesses, including mental disorders, drug addiction, abnormal personality, and poorly controlled schizophrenia;
* (3) Regularly take sedative and sleeping drugs or central nervous system stimulants
* (4) Major physical diseases, including cancer, poorly controlled diabetes, hypertension and thyroid disease, immune rheumatism, heart failure, chronic obstructive pulmonary disease, liver cirrhosis, and chronic kidney disease stages IV and V

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Laser Doppler blood flow analysis (perfusion unit (PU)) | Baseline
  It is a technique for monitoring microvascular perfusion by PeriFlux System 5000 (Perimed, Stockholm, Sweden). The light source can penetrate tissues and thus can measure blood perfusion without invasive procedures. The microvascular perfusion situation is immediate results and can be used to quantify the degree of skin damage. Its unit is perfusion unit (PU).
Laser Doppler blood flow analysis (perfusion unit (PU)) | 12 weeks
  It is a technique for monitoring microvascular perfusion by PeriFlux System 5000 (Perimed, Stockholm, Sweden). The light source can penetrate tissues and thus can measure blood perfusion without invasive procedures. The microvascular perfusion situation is immediate results and can be used to quantify the degree of skin damage. Its unit is perfusion unit (PU).
Laser Doppler blood flow analysis (perfusion unit (PU)) | 26 weeks
  It is a technique for monitoring microvascular perfusion by PeriFlux System 5000 (Perimed, Stockholm, Sweden). The light source can penetrate tissues and thus can measure blood perfusion without invasive procedures. The microvascular perfusion situation is immediate results and can be used to quantify the degree of skin damage. Its unit is perfusion unit (PU).

SECONDARY OUTCOMES:
Hydration | Baseline
  The skin multi-functional detection system measures the skin's water content to detect whether the skin is too dry.
Hydration | 12 weeks
  The skin multi-functional detection system measures the skin's water content to detect whether the skin is too dry.
Hydration | 26 weeks
  The skin multi-functional detection system measures the skin's water content to detect whether the skin is too dry.
Transepidermal water loss | Baseline
  Use the skin multifunctional detection system to measure the skin water loss state to understand the skin health.
Transepidermal water loss | 12 weeks
  Use the skin multifunctional detection system to measure the skin water loss state to understand the skin health.
Transepidermal water loss | 26 weeks
  Use the skin multifunctional detection system to measure the skin water loss state to understand the skin health.
Sebum | Baseline
  The measuring principle is to use a photometer to measure the oil point transmittance to determine the size of the oil point and detect the skin oil content.
Sebum | 12 weeks
  The measuring principle is to use a photometer to measure the oil point transmittance to determine the size of the oil point and detect the skin oil content.
Sebum | 26 weeks
  The measuring principle is to use a photometer to measure the oil point transmittance to determine the size of the oil point and detect the skin oil content.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Investigators do not plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Yu WT, Yu HS, Wu CS, Lee CH, Cheng YC, Lin WT, Chen GS, Lan CC. Noninvasive cutaneous blood flow as a response predictor for visible light therapy on segmental vitiligo: a prospective pilot study. Br J Dermatol. 2011 Apr;164(4):759-64. doi: 10.1111/j.1365-2133.2010.10148.x. PMID 21087230
- [Background] Yang SY, Lan CC. Acquired Port-wine Stain with Local Heat. Acta Derm Venereol. 2016 Feb;96(2):274-5. doi: 10.2340/00015555-2193. No abstract available. PMID 26123172